CLINICAL TRIAL: NCT02514720
Title: Influence of Nicotine Metabolism Ratio on [11C]-(+)-PHNO PET Binding in Tobacco Smokers
Brief Title: Nicotine Metabolizers and [11C]-(+)-PHNO
Acronym: MET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Bernard Le Foll, Head of the Translational Addiction Research Laboratory, Centre for Addiction and Mental Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 111/2014
Record Dates: First submitted 2015-07-30; First posted 2015-08-04 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2017-06

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tobacco Products

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fast Nicotine Metabolizers (Other): Those in the upper tertile of NMR for cigarette/nicotine metabolism.
  Interventions: Other: cigarette
- Slow Nicotine Metabolizers (Other): Those in the lower tertile of NMR for cigarette/nicotine metabolism
  Interventions: Other: cigarette

INTERVENTIONS:
Other: cigarette — Participants will be allowed to smoke a cigarette prior to a PET scan and be abstinent from smoking prior to the other PET scan

SUMMARY:
The purpose of this study is to investigate the effects of nicotine metabolism on occupancy of [11C]-(+)-PHNO to DA 2/3 receptors in different brain areas during periods of abstinence and smoking during an abstinence. This will be a Positron Emission Tomography (PET) study and the radiotracer [11C]-(+)-PHNO (11C]-( + )-4-propyl- 3,4,4a,5,6,10b-hexahydro-2H-naphtho[1,2-b][1,4]oxazin-9-ol) will be used.

DETAILED DESCRIPTION:
The participants will undergo a PET scan after approximately 48 hours abstinence (to ensure total elimination of nicotine in both FMs and SMs) and then approximately >5 hours later may have a second PET scan after smoking their preferred cigarette (approximately 1 hour before). It is possible that these two scans may also occur on separate days. All subjects will provide a urine sample for (1) drug toxicology, (2) pregnancy test (in females) and (3) Total Nicotine Equivalents (TNE: a measure of total consumption unaltered by rate of nicotine metabolism). There will one blood draw taken before and one after each PET scan (about 20mls in total) to measure nicotine and COT levels (to assess abstinence) as well as kinetics of nicotine delivery. Participants will be given questionnaires prior to, or during, and/or after one or both of the PET scans to determine differences between abstinence and smoking on subjective measures..

ELIGIBILITY:
Inclusion Criteria:

* Males and females of any ethnic origin 18 years of age or older.
* No previous use of medication for smoking cessation in previous month-
* Non-treatment seeker
* Either SMs or FMs by NMR

Exclusion Criteria:

* DSM-IV diagnosis of other drug dependences
* Any medical condition requiring immediate investigation or treatment
* Pregnancy tested by urine or lactation by self-report
* Current diagnosis of any Axis I psychiatric disorder
* Regular use of any therapeutic or recreational psychoactive drug use that may interfere with PET scanning
* Exposure to radiation in the last 12 months exceding permissible limit for participants participating in research
* Current use of medication that may interfere with [11C]-(+)-PHNO
* Metal implants or paramagnetic objects within the body which may interfere with the MRI
* Claustrophobia or a history of panic attacks
* Having any clinical condition, drug sensitivity, or prior therapy which, in the investigator's opinion, makes the participant unsuitable for the study
* Current use of antidepressants that may inhibit CYP2A6 or impact response to nicotine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Occupancy of D2/3 receptors by [11C]-(+)-PHNO | 2 weeks
  Fast and slow nicotine metabolizers will have PET scans and occupancy of dopamine receptors will be measured using a PET scanner.

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Le Foll, MD, PHD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Di Ciano P, Tyndale RF, Mansouri E, Hendershot CS, Wilson AA, Lagzdins D, Houle S, Boileau I, Le Foll B. Influence of Nicotine Metabolism Ratio on [11C]-(+)-PHNO PET Binding in Tobacco Smokers. Int J Neuropsychopharmacol. 2018 Jun 1;21(6):503-512. doi: 10.1093/ijnp/pyx119. PMID 29346545
- See also: Published data may be found at site above and PMID 29346545 — https://www.ncbi.nlm.nih.gov/pubmed/29346545